CLINICAL TRIAL: NCT05641584
Title: The Effect of Preoperative Monocyte/HDL Ratio on Postoperative Mortality and Morbidity in Patients Undergoing Aortic Valve Replacement for Aortic Stenosis-Retrospective Study
Brief Title: Is Monocyte/HDL Ratio a Predictor of Mortality in Aortic Valve Surgery
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Tuğba Yücel,MD, Principal Investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: 2022/155
Record Dates: First submitted 2022-11-29; First posted 2022-12-07 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Inflammation; Aortic Valve Stenosis; HDL
MeSH Terms: conditions — Inflammation; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: retrospective data review study — Patient information will be scanned retrospectively from the computer environment and patient cards. No intervention will be made to the patients.

SUMMARY:
In this study, the investigators aimed to determine whether the preoperative Monocyte/HDL ratio would be a predictor of postoperative mortality and morbidity in patients who underwent aortic valve replacement due to aortic stenosis.

DETAILED DESCRIPTION:
Inflammation is causally associated with both coronary artery disease and aortic stenosis. Although aortic stenosis is considered a static degenerative and calcific process, recent evidence has shown the opposite. The role of inflammation in the pathogenesis of AS It will be investigated that mortality may be associated with increased inflammation in patients treated with AVR.

Adult patients (aged ≥18 years) with ASA II-IV who underwent elective aortic valve replacement under cardiopulmonary bypass (CPB) due to aortic stenosis in our clinic between January 1, 2010 and March 31, 2022, will be included in the study by retrospectively scanned from the computer system and patient cards. The exclusion criteria from the study are as follows; those with signs of acute infection, those with autoimmune disease, those with severe renal (serum creatinine >2.0 mg/dl) disease, those with severe hepatic disease, those with suspected malignancy.

Demographic characteristics of patients (age, gender, body mass index, diabetes mellitus, hypertension, chronic kidney disease-failure, peripheral vascular disease, smoking history, hyperlipidemia, atrial fibrillation history, left ventricular ejection fraction, coronary artery disease history, Cabg history) Europe Cardiac Operative Risk Assessment System II (EuroSCORE), Systemic Immune-Inflammatory Index (SII), APACHE II, SOFA Score, NYHA III/IV values, drugs used (ASA, oral anticoagulants, beta blocker, statin, ACE inh., ARB) , preoperative glucose, HbA1c, urea, creatinine, total cholesterol, LDL, HDL, triglyceride, hemoglobin, hematocrit, platelet, WBC, neutrophil, lymphocyte, monocytes, monocyte/HDL ratio, CRP, preoperative and postoperative EF and PAB values, ICU admission duration, duration of invasive mechanical ventilation, type of discharge, amount of ES replaced will be recorded. Operation time, cardiopulmonary bypass (extracorporeal circulation) time, cross clamp time, inotropic and vasopressor requirements will be recorded)

ELIGIBILITY:
Inclusion Criteria:

be over the age of 18, ASA II-IV Patients scheduled for cardiac surgery due to on-pomp aortic valve replacement

Exclusion Criteria:

emergency operations, off pump)pumpless surgery, revision (repetitive) operations, those with signs of acute infection, those with autoimmune disease, those with severe renal (serum creatinine >2.0 mg/dl) disease, those with severe hepatic disease, those with suspected malignancy, patients where data variables cannot be saved due to technical problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in the study Adult patients (aged ≥18 years) with ASA II-IV who underwent elective aortic valve replacement under Cardiopulmonary bypass (CPB) for aortic stenosis in our clinic between January 1, 2010 and March 31, 2022, were retrospectively scanned from the computer system and patient cards, and included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
mortality | 6 month
  The investigators aimed to determine whether the preoperative Monocyte/HDL ratio would be a predictor of postoperative mortality in patients who underwent aortic valve replacement due to aortic stenosis.
morbidity | 6 month
  The investigators aimed to determine whether the preoperative Monocyte/HDL ratio would be a predictor of postoperative mortality and The investigators aimed to determine whether the preoperative Monocyte/HDL ratio would be a predictor of postoperative mortality and morbidity in patients who underwent aortic valve replacement due to aortic stenosis. in patients who underwent aortic valve replacement due to aortic stenosis.

SECONDARY OUTCOMES:
Inflammation | 6 month
  Inflammation is causally associated with both coronary artery disease and aortic stenosis. Although aortic stenosis is considered a static degenerative and calcific process, recent evidence has shown the opposite. The role of inflammation in the pathogenesis of AS It will be investigated that mortality may be associated with increased inflammation in patients treated with AVR.

CONTACTS AND LOCATIONS:
Overall Officials: tuğba yücel, md, Principal Investigator — Bakirkoy Dr Sadi Konuk Traning Hospital
Locations (1):
- ISTANBUL Bakırkoy Dr. Sadi Konuk Training and Research Hospital,, Istanbul, Bakırköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided